CLINICAL TRIAL: NCT05702021
Title: Implementing Contingency Management for Stimulant Use in Specialty Addiction Treatment Organizations (Center for Dissemination and Implementation Science at Stanford, Research Component #2)
Brief Title: Implementing Contingency Management for Stimulant Use in Specialty Addiction Treatment Organizations
Acronym: MIMIC2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Stanford University (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Sara Becker, Alice Hamilton Professor of Psychiatry, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00217287; P50DA054072 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-01-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stimulant Use (Diagnosis)
Keywords: Stimulants; Contingency management; Opioid Use Disorder; Implementation science; Behavior change
MeSH Terms: conditions — Disease; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Stepped-wedge trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be exported from electronic medical records. Data analysts will not know who was receiving the intervention at what time point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Science of Service Laboratory implementation strategy (Experimental): The Science of Service Laboratory implementation strategy consists of: didactic training (contingency management workshops; monthly contingency management coaching calls), performance feedback (practice sessions and electronic medical record feedback); and facilitation (monthly facilitation calls).
  Interventions: Behavioral: Science to Service Laboratory
- Stepped wedge comparator (No Intervention): Our hybrid trial uses a unidirectional crossover stepped wedge design. All sites cross over in the same direction from usual care to intervention. All sites therefore act as their own comparison prior to the sequential roll-out of the implementation strategy.

INTERVENTIONS:
Behavioral: Science to Service Laboratory — The Science of Service Laboratory implementation strategy consists of: didactic training (contingency management workshops; monthly contingency management coaching calls), performance feedback (practice sessions and electronic medical record feedback); and facilitation (monthly facilitation calls).
  Arms: Science of Service Laboratory implementation strategy

SUMMARY:
Stimulants constitute a new and deadly fourth wave of the opioid epidemic. Contingency management is the most effective intervention for stimulant use and is an evidence-based adjunct to medication for opioid use disorder. Yet, uptake of contingency management in opioid treatment programs that provide medication for opioid use disorder remains low; in fact, access to contingency management is arguably one of the greatest research-to-practice gaps in the addiction treatment services field. The goal of this study is to conduct a type III hybrid effectiveness-implementation trial to evaluate a multi-level implementation strategy, the Science of Service Laboratory, to install contingency management for stimulant use in opioid treatment programs. The Science of Service Laboratory has three core components: didactic training, performance feedback, and external facilitation.

Utilizing a stepped wedge design, a regional cohort of 10 public sector opioid treatment programs will be randomized to receive Science of Service Laboratory at five distinct time points. At six intervals, each of the 10 opioid treatment programs will provide de-identified electronic medical record data from all available patient charts on contingency management delivery and patient outcomes. Staff from each opioid treatment program will provide feedback on contextual determinants influencing implementation. This study will rigorously evaluate whether a multi-level implementation strategy developed by one of the longest-standing national intermediary purveyor organizations-the SAMHSA Technology Transfer Centers, will improve both implementation and patient outcomes.

DETAILED DESCRIPTION:
Stimulant use among persons with opioid use disorder is associated with an array of serious consequences. Among those with opioid use disorder, stimulant use has been associated with more persistent opioid use; higher risk of HIV infection; higher levels of family, medical, legal, and vocational problems; and increased risk of fatal overdose. Contingency management is an evidence-based intervention for stimulant use and an evidence-based adjunct to medication for opioid use disorders. Medication for opioid use disorder is the first-line, evidence-based treatment for opioid use disorder, but does not specifically reduce stimulant use, and there are not yet efficacious medications for stimulant addiction. Moreover, individuals who continue to use stimulants while receiving medication for opioid use disorder have worse treatment response in terms of both retention and abstinence from opioids. Contingency management targets stimulant use via reinforcing incentives for attaining abstinence. Despite an abundance of research evidence, contingency management uptake in opioid treatment programs remains low due to barriers at both the provider- and organizational-levels. Effectively addressing the contingency management evidence-to-practice gap could advance both the field of implementation science and the quality of care in specialty addiction treatment settings. This project evaluates a multi-level implementation strategy, the Science to Service Laboratory, to install contingency management for stimulant use in opioid treatment programs. The Science of Service Laboratory employs three core components: didactic training; performance feedback; and external facilitation.

Utilizing a fully powered type III hybrid effectiveness-implementation trial with a stepped wedge design, we will randomize a cohort of 10 public sector opioid treatment programs in New England to receive the Science of Service Laboratory at five time points. Data collection will leverage multiple sources. At six intervals, each of the 10 opioid treatment programs will extract de-identified electronic medical record data on contingency management implementation and patient outcomes. In addition, opioid treatment program staff will report on contextual determinants of implementation. Results will evaluate whether a multi-level implementation strategy initially developed by one of the longest-standing intermediary purveyor organizations (SAMHSA Technology Transfer Centers), will improve implementation and patient outcomes. In addition, the project will ensure equitable service provision to diverse, high-risk patients while advancing implementation science via specification and evaluation of contextual determinants.

The Specific Aims and corresponding hypotheses are:

Specific Aim 1: To test the effectiveness of the Science of Service Laboratory on implementation outcomes, including contingency management Reach, Adoption, and Implementation.

Specific Aim 2: To test the effectiveness of the Science of Service Laboratory on patient outcomes, including: Stimulant Abstinence and Treatment Retention.

ELIGIBILITY:
* Opioid Treatment Program Counselors:

  * Inclusion criteria: 1) provide ongoing psychosocial support to medication for opioid use disorder patients (e.g., intake sessions, individual counseling, and/or group counseling sessions), and 2) have an active caseload
  * Exclusion criteria: Younger than 18 years of age, unable to provide informed consent
* Persons on Medication for Opioid Use Disorder [Not recruited, via electronic medical records only]

  * Inclusion criteria: must be newly initiated on medication for opioid use disorders (within the past 30 days) and have concurrent stimulant use (indicated by self-report of past 30-day stimulant use or positive toxicology screen within 30 days).
  * Exclusion criteria: Younger than 18 years of age, Does not have electronic medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in percent of patients receiving contingency management from pre-implementation to post-implementation | 10 months
  This is an implementation outcome capturing Reach and is extracted from electronic medical records. This is a patient-level measure of the change in the percent of newly inducted patients with a history of stimulant use who are documented as having received 1 or more contingency management sessions from pre-implementation to post-implementation.
Change in percent of counselors delivering contingency management from pre-implementation to post-implementation | 10 months
  This is an implementation outcome capturing Adoption and is extracted from electronic medical records. This is a provider-level measure of the change in percent of counselors at each program who are documented as having delivered 1 or more contingency management sessions from pre-implementation to post-implementation.

SECONDARY OUTCOMES:
Change in the percent of toxicology screens negative for stimulants | 10 months
  This is a patient-level outcome measuring Stimulant Abstinence and is extracted from electronic medical records. This measures the change in percent of toxicology screens that are negative for stimulants from pre-implementation to post-implementation.
Change in number of contingency management sessions | 10 months
  This is a patient-level outcome measuring Contingency Management Treatment Retention and is extracted from electronic medical records. This measures the change in the number of contingency management sessions received per patient from pre-implementation to post-implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Becker, Principal Investigator — Northwestern University
Locations (10):
- United States (10):
  - Lawndale Christian Health Center, Chicago, Illinois
  - Healthcare Alternative Systems NEXA-MAR, Chicago, Illinois
  - Community Outreach Intervention Projects Southside Mobile Van, Chicago, Illinois
  - Family Guidance Centers Chicago Ave., Chicago, Illinois
  - Addiction Recovery Institute, Pawtucket, Rhode Island
  - CODAC Pawtucket, Pawtucket, Rhode Island
  - Providence Comprehensive Treatment Center, Providence, Rhode Island
  - VICTA, Providence, Rhode Island
  - CODAC Providence, Providence, Rhode Island
  - Woonsocket Comprehensive Treatment Center, Woonsocket, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
This study protocol is embedded within a Center of Excellence funded by the National Institute on Drug Abuse. In coordination with other center project components, the study protocol and statistical analysis plan for primary outcomes will be submitted for publication to either an addiction (e.g., Addiction, Journal of Substance Abuse Treatment) or implementation science (e.g., Implementation Science, Implementation Science: Research and Practice) journal. Additional data (analytic code, participant-level data) can be requested from the Principal Investigator. Analysis files will be constructed from the electronic data and will be stripped of identifying information. Specifically, participants will be identified with a numeric identifier that is not related to any element of their personal identifying information. No names, addresses, telephone numbers, email addresses, medical record numbers, etc. will be retained in the de-identified files.
Supporting Information: Study Protocol, SAP
Time Frame: Protocol will be submitted for publication in coordination with other project components, with a target submission date in 2023. Analytic code and participant-level data will be made ready for distribution within 12 months of study completion.
Access Criteria: Data will only be shared with external investigators when a data use agreement (DUA) is executed between Northwestern University and the requester's institution. The DUA will specify the requested data elements (each of which must be justified), the specific research question, the timeline for the project, and schedule for data destruction.

REFERENCES:
- [Derived] Becker SJ, DiClemente-Bosco K, Scott K, Janssen T, Salino SM, Hasan FN, Yap KR, Garner BR. Implementing contingency management for stimulant use in opioid treatment programs: protocol of a type III hybrid effectiveness-stepped-wedge trial. Implement Sci. 2023 Sep 13;18(1):41. doi: 10.1186/s13012-023-01297-w. PMID 37705093